CLINICAL TRIAL: NCT04943081
Title: The Effect of Percutaneous Nephrolithotomy on the Estimated Glomerular Filtration Rate in Patients With Stage 2-4 Chronic Kidney Disease
Brief Title: Percutaneous Nephrolithotomy in Patients With Stage 2-4 Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelghany Allam, Assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCNL in chronic kidney disease
Record Dates: First submitted 2021-06-18; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Percutaneous Nephrolithotomy
MeSH Terms: interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Intervention Model Description: Adult patients with age group ≥ 18 years old with renal stones candidate for PCNL with pre-operative estimated GFR less than 90 ml/min/1.7 m2 and ≥ 15 ml/min/1.7 m2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Case group (Experimental): Adult patients with age group ≥ 18 years old with renal stones candidate for PCNL with pre-operative estimated GFR less than 90 ml/min/1.7 m2 and ≥ 15 ml/min/1.7 m2.
  Interventions: Procedure: Percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: Percutaneous nephrolithotomy — Percutaneous nephrolithotomy (PCNL) is a technique used to remove complex renal stones, or stones resistant to shockwave lithotripsy. A tube is placed through the incision in the kidney, under X-ray guidance, and renal stones are extracted by using nephroscope

SUMMARY:
The study aims to evaluate the effect of percutaneous nephrolithotomy (PCNL) on estimated glomerular filtration rate (eGFR) in patients with stage 2-4 chronic kidney disease

DETAILED DESCRIPTION:
Nephrolithiasis affects an estimated 5-10% of the general population, and this percentage continues to rise. It has a prevalence of 1.7% to 18% in patients with chronic kidney disease (CKD), and nephrolithiasis-related CKD contributed to 3.2% of the total patients who started maintenance dialysis therapy.

The etiology of renal insufficiency in patients with nephrolithiasis is multifactorial and includes renal obstruction, recurrent urinary tract infections, frequent surgical interventions and coexisting medical disease.

According to National kidney foundation, chronic kidney disease is classified into 5 stages as follows:

Stage 1: Kidney damage with normal or elevated GFR < 90 ml/min/1.7 m2 Stage 2: Kidney damage with mildly decreased GFR 60-89 ml/min/1.7 m2 Stage 3: Moderately decreased GFR 30-59 ml/min/1.7 m2 Stage 4: Severely decreased GFR 15-29 ml/min/1.7 m2 Stage 5: Kidney Failure GFR>15 ml/min/1.7 m2 Management of nephrolithiasis in patients with CKD is often difficult. Options for preserving kidney function include watchful waiting, shockwave lithotripsy (SWL), an endourologic approach (Percutaneous nephrolithotomy or retrograde intra-renal surgery), laparoscopic surgery or conventional open surgery.

Percutaneous nephrolithotomy (PCNL) is considered as the gold standard intervention for large burden and complex renal stone disease and is associated with the highest stone free rates (SFRs). However, potentially significant complications include bleeding, sepsis, pleural and visceral injury. Therefore, the optimal management plan needs to be tailored to individual patient.

Serum creatinine level has been used as a crude index of renal function in studies of patients with CKD, but it is not reliable. The glomerular filtration rate (GFR) should be used instead. GFR is the most accurate way to give health providers an estimate of functioning renal mass. Estimating GFR with the use of prediction equations is cost effective.

In this study, we will prospectively evaluate the effect of percutaneous nephrolithotomy on the estimated glomerular filtration rate in Patients With Stage 2-4 chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with age group ≥ 18 years old with renal stones candidate for PCNL with pre-operative estimated GFR less than 90 ml/min/1.7 m2 and ≥ 15 ml/min/1.7 m2

Exclusion Criteria:

* Patients with chronic renal failure on regular dialysis.
* Patients with bleeding diathesis.
* Patients who are unfit for surgery.
* Pregnancy
* Patients who are refusing the participation in our study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Estimation of GFR for all patients pre-operative | 1 day pre-operative
  Estimation of GFR for all patients pre-operative by using body surface area based-Cockcroft-Gault formula (CG/ BSA).
  Body surface area based Cockcroft-Gault formula (CG/ BSA) = [(140- age) x weight in kilograms x (0.85 if female)] / (72 x serum creatinine in mg/dl).
  This formula expects weight to be measured in kilograms and creatinine to be measured in mg/dl.
Estimation of GFR for all patients three months post-operative | 3 months post-operative
  Estimation of GFR for all patients three months post-operative by using body surface area based-Cockcroft-Gault formula (CG/ BSA).
  Body surface area based Cockcroft-Gault formula (CG/ BSA) = [(140- age) x weight in kilograms x (0.85 if female)] / (72 x serum creatinine in mg/dl).
  This formula expects weight to be measured in kilograms and creatinine to be measured in mg/dl.

CONTACTS AND LOCATIONS:
Overall Officials: Adel Kurkar, Study Director — Assiut University; Ahmed Moeen, Study Director — Assiut University; Amr Abo-Faddan, Study Director — Assiut University

REFERENCES:
- [Background] Edvardsson VO, Indridason OS, Haraldsson G, Kjartansson O, Palsson R. Temporal trends in the incidence of kidney stone disease. Kidney Int. 2013 Jan;83(1):146-52. doi: 10.1038/ki.2012.320. Epub 2012 Sep 19. PMID 22992468
- [Background] Gupta M, Bolton DM, Gupta PN, Stoller ML. Improved renal function following aggressive treatment of urolithiasis and concurrent mild to moderate renal insufficiency. J Urol. 1994 Oct;152(4):1086-90. doi: 10.1016/s0022-5347(17)32509-0. PMID 8072069
- [Background] Jungers P, Joly D, Barbey F, Choukroun G, Daudon M. ESRD caused by nephrolithiasis: prevalence, mechanisms, and prevention. Am J Kidney Dis. 2004 Nov;44(5):799-805. PMID 15492945
- [Background] Gambaro G, Favaro S, D'Angelo A. Risk for renal failure in nephrolithiasis. Am J Kidney Dis. 2001 Feb;37(2):233-43. doi: 10.1053/ajkd.2001.21285. PMID 11157364
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Gopalakrishnan G, Prasad GS. Management of urolithiasis with chronic renal failure. Curr Opin Urol. 2007 Mar;17(2):132-5. doi: 10.1097/MOU.0b013e328028fdfb. PMID 17285024
- [Background] Jones P, Aboumarzouk OM, Rai BP, Somani BK. Percutaneous Nephrolithotomy for Stones in Solitary Kidney: Evidence From a Systematic Review. Urology. 2017 May;103:12-18. doi: 10.1016/j.urology.2016.10.022. Epub 2016 Nov 14. PMID 27856206